CLINICAL TRIAL: NCT05264805
Title: A Randomized Controlled Trial of Port Site Subcutaneous Injection of Bupivacaine to Determine the Effectiveness of Postoperative Pain Relief After Laparoscopic Cholecystectomy
Brief Title: Effectiveness of Port Site Bupivacaine Injection in Postoperative Pain Reduction After Lap. Chole
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamdard University (Other)
Responsible Party: Principal Investigator, Dr. Nida Shahid, Assistant Professor, Hamdard University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N0333
Record Dates: First submitted 2022-02-04; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Pain, Postoperative
Keywords: #Post operative pain; #laparoscopic cholecystectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Group A:
  Study group: Patient receiving intervention i.e 20ml of 0.25% buvivacaine infiltration at laparoscopic port site.
  Group B:
  Control group: no intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine group (Experimental): Patient receiving 20ml of inj. 0.25% Bupivacaine at laparoscopic port site
  Interventions: Drug: 0.25% Bupivacaine
- Placebo group (No Intervention): No drug infiltration at laparoscopic port site

INTERVENTIONS:
Drug: 0.25% Bupivacaine — 20ml of 0.25% Bupivacaine subcutaneous infiltration at port site wound.
  Other Names: Bupivacain
  Arms: Bupivacaine group

SUMMARY:
To determine the effectiveness of port site bupivacaine infiltration in postoperative pain reduction after laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
The study is being done to determine the effectiveness of port site bupivacaine infiltration in postoperative pain reduction after laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both the gender of age >18 years and <45years
2. Patients undergoing elective laparoscopic cholecystectomy under general anesthesia.
3. Patients with A.S.A grade I and II.

Exclusion Criteria:

1. Patients with known allergic reactions to local anesthetics.
2. Patients converted to open procedure.
3. Patients developing intra-operative complications.
4. Patients undergoing for laparoscopic cholecystectomy for acute cholecystitis.
5. Patients with obesity and chronic illness.
6. Patients with history of opioids, steroids, NSAIDs and alcohol use.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 166 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Post laparoscopic port site pain assessment | Pain assessment from 0hour (patient received in recovery room) till 12hours postoperatively at interval of 3hours i.e. 0,3,6,9,12 hour
  Pain assessment by "Visual Analog Scoring system" scoring from 0 to 10, where 0 means no pain and 10 means worst possible, unbearable excruciating pain.